CLINICAL TRIAL: NCT02253823
Title: A Single Center, Open-Label, Randomised, Parallel, Multiple Dose Comparison of the Effect of Tipranavir 500 mg and Ritonavir 100 mg or Tipranavir 750 mg and Ritonavir 200 mg, Administered Daily on 3 Non-Consecutive Days and Twice Daily for 7 Days, on the Pharmacokinetic Characteristics of Efavirenz (Sustiva®) 600 mg a Day in Healthy Adult Volunteers
Brief Title: Multiple Dose Comparison of the Effect of Two Dose Combinations of Tipranavir/Ritonavir (TPV/RTV), on the Pharmacokinetic Characteristics of Efavirenz (Sustiva®) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1182.41
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (2):
- TPV+RTV - low dose (Experimental)
  Interventions: Drug: EFV; Drug: TPV/RTV - low dose
- TPV+RTV - high dose (Experimental)
  Interventions: Drug: EFV; Drug: TPV/RTV - high dose

INTERVENTIONS:
Drug: EFV
Drug: TPV/RTV - low dose
  Arms: TPV+RTV - low dose
Drug: TPV/RTV - high dose
  Arms: TPV+RTV - high dose

SUMMARY:
The objective of this study was to characterize the effects of two dose combinations of tipranavir/ritonavir (TPV 500 mg/RTV 100 mg and TPV 750 mg/RTV 200 mg), administered daily and BID, on the pharmacokinetics of efavirenz (EFV), 600 mg daily

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to give written informed consent in accordance with institutional and federal guidelines and to comply with the investigational nature of the study and the related requirements
* Healthy males or females between 18 and 60 years of age inclusive
* Ability to swallow numerous large capsules without difficulty
* Reasonable probability for completion of the study
* A Body Mass Index (BMI) between 18 and 35 kg/m2
* Acceptable laboratory values that indicate adequate baseline organ function are required at the time of screening. Laboratory values are considered to be acceptable if severity ≤ Grade 1 based on the Adult AIDS Clinical Trial Group (ACTG) Division of Acquired Immunodeficiency Syndrome (of the National Institute of Allergy and Infectious Diseases / National Institutes of Health) (DAIDS) Grading Scale. All abnormal laboratory values > Grade 1 (e.g., creatine phosphokinase (CPK), amylase, triglycerides) are subject to approval by the Boehringer Ingelheim Pharmaceuticals, Inc. (BIPI) clinical monitor
* Acceptable medical history, physical examination, ECG, and Chest X-ray are required prior to entering the study
* Willingness to abstain from alcohol for 48 hours prior to Study Day 0 and abstain from alcohol for the duration of the study. In addition, Cabernet Sauvignon must not have been ingested within 15 days prior to Day 0 (Visit 2)
* Willingness to abstain from ingesting grapefruit and grapefruit juice within 15 days of Day 0, Visit 2 and for the duration of the study
* Willingness to abstain from ingesting Seville oranges, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc.) within 72 hours of PK sampling days [Visit 3 (Days 1-6), Visit 4 (Days 12-15), Visit 5 (Days 20-21 and Visit 6 (Day 22)]
* Willingness to abstain from use of tobacco products for the duration of the study
* Urine drug screen negative for illegal non-prescription drugs
* Negative HIV serology
* Negative for Hepatitis B surface antigen and Hepatitis C

Exclusion Criteria:

* Female subjects who are of reproductive potential who:

  * Have a positive serum B-human chronic gonadotropin (HCG) at Visit 1 or,
  * Have not been using a barrier contraceptive method for at least 3 months prior to Visit 3 (Day 1), or
  * Are not willing to use a reliable method of double-barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam) during the trial and 30 days after completion/termination or,
  * Are breast-feeding
* Participation in another trial with an investigational medicine for 30 days prior to Day 0 (Visit 2)
* Use of any known enzyme altering drug (such as phenothiazines, cimetidine, barbiturates, ketoconazole, fluconazole, rifampin, steroids, and herbal medications within 30 days prior to Day 0 (Visit 2) or during the trial
* Ingestion of grapefruit, grapefruit juice, and Cabernet Sauvignon within 15 days prior to Day 0 (Visit 2)
* Ingestion of Seville oranges, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc.) within 72 hours of pharmacokinetics (PK) sampling days [Visit 3 (Days 1-6), Visit 4 (Days 12-15), Visit 5 (Days 20-21 and Visit 6 (Day 22)]
* Administration of antibiotics within 10 days prior to Day 0 (Visit 2) or during the trial
* Inability to comply with investigator's instructions
* History of central nervous system (CNS), gastrointestinal, hepatic, or renal disorders within the past 60 days. Subjects were excluded for these disorders greater than sixty days, if in the opinion of the investigator, the subject did not qualify as a healthy volunteer
* History of alcohol abuse
* Excessive cigarettes smoking defined as greater than 10 cigarettes per day
* Blood or plasma donations within 30 days prior to Day 0 (Visit 2)
* Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >90 beats/min. For subjects with a resting heart rate below 50, due to high fitness level, the investigator could discuss exclusion with medical monitor on a case-by-case basis
* Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering tipranavir, ritonavir or efavirenz to the subject
* Subjects who have an acute illness within 2 weeks prior to Day 0 (Visit 2).
* Subjects who are taking any over-the-counter drug within 7 days prior to Day 0, (Visit 2) or are taking any prescription drug that, in the opinion of the investigator in consultation with the BIPI clinical monitor and pharmacokineticist, might interfere with either the absorption, distribution or metabolism of the test substances
* Subjects suffering from active forms of depression
* Subjects that had a history of suicidal ideations
* Known hypersensitivity to tipranavir, ritonavir, or efavirenz

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2001-12; Primary Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration
AUC 0-12 (Area under the plasma concentration time curve from 0-12 hours) | up to 12 hours after drug administration
Cp12h (observed drug concentration in plasma at 12 hours) | up to 12 hours after drug administration
AUC 0-24 (Area under the plasma concentration time curve from 0-24 hours) | up to 24 hours after drug administration
Cp24h (observed drug concentration in plasma at 24 hours) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 24 hours after drug administration
V (Volume of distribution) | up to 24 hours after drug administration
Tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 24 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 24 hours after drug administration
Number of subjects with adverse events | up to 43 days
Number of subjects with abnormal changes in laboratory parameters | up to 43 days